CLINICAL TRIAL: NCT00530803
Title: The Efficacy of the Eutectic Mixture of Local Anesthetics (EMLA) Cream Versus the Synera Patch for Pain Reduction During Venipuncture in Children
Brief Title: The Efficacy of EMLA Cream vs. Synera Patch for Pain Reduction During Venipuncture in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 07-06-159
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-07

CONDITIONS: Pain; Needle Phobia
Keywords: EMLA; venipuncture; children; Synera patch; pediatric; Lidocaine/prilocaine
MeSH Terms: conditions — Pain | interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EMLA Cream (Active Comparator): Participants will have a dose of EMLA Cream applied to the venipuncture site 1 hour before the procedure. Dosage based on age and weight: 4-6 years old and heavier than 10kg will receive 10g of EMLA; 7-12 years old and more than 20kg will receive 20g of EMLA.
  Interventions: Drug: EMLA Cream
- Synera Patch (Active Comparator): Participants will have a Synera Patch applied to the venipuncture site 20 minutes prior to the procedure.
  Interventions: Combination Product: Synera Patch

INTERVENTIONS:
Drug: EMLA Cream — 60 minutes x1
  Other Names: Lidocaine/prilocaine cream
  Arms: EMLA Cream
Combination Product: Synera Patch — 20 minutes x1
  Other Names: Lidocaine/tetracaine patch
  Arms: Synera Patch

SUMMARY:
This study compares the efficacy of the Synera patch with Eutectic Mixture of Local Anesthetics (EMLA) as a topical anesthetic for venipuncture in pediatric patients.

DETAILED DESCRIPTION:
Venipunctures are common and necessary components of pediatric health care. Unfortunately, many children have "needle phobia" and even a simple procedure, such as a venipuncture, can cause significant stress and anxiety to the patient and the parents involved. Studies have shown that needles are the worst part of hospital/healthcare related visits for children.

The Synera patch uses a controlled heating system to transcutaneously deliver a lidocaine/tetracaine mixture for analgesic effect. No published studies compare the efficacy of the Synera patch with other topical anesthetics in children. The objective of this study is to compare the efficacy of the Synera patch applied for 20 minutes with the efficacy of EMLA Cream applied for 60 minutes in reducing pain associated with venipunctures in children.

Patients, 4-12 years old children requiring venipunctures in clinics, were randomized to receive Synera for 20 minutes or EMLA for 60 minutes. A blinded observer recorded pain scores using a numerical rating scale (NRS). Child and parent assessed pain with the Wong-Baker FACES Scale and the NRS, respectively. The primary outcome was the number of subjects reporting "no pain". Secondary outcomes were parent and observer measures of the child's pain and the presence of skin reactions.

ELIGIBILITY:
Inclusion Criteria:

* Children in outpatient clinics requiring venipuncture for medical care
* Ages 4-12 years old
* The ability to demonstrate proper understanding of the Wong-Baker FACES Pain Ranking Scale
* Parents of enrolled children need to be present during the procedure and be willing to rate their child's pain

Exclusion Criteria:

* Damaged or inflamed skin at the designated application site
* Known sensitivity to components of Synera or EMLA (lidocaine, tetracaine, or local anesthetics of the amide or ester type, Para Aminobenzoic (PABA) derivatives)
* Contraindications to SYnera or EMLA use (Severe hepatic disease, history of drug-induced methemoglobinemia, taking Class 1 antiarrhythmics)
* Use of analgesics during the past 24 hours

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine C Skae, MD, Principal Investigator — Children's Hospital at Montefiore
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States

REFERENCES:
- [Background] Arts SE, Abu-Saad HH, Champion GD, Crawford MR, Fisher RJ, Juniper KH, Ziegler JB. Age-related response to lidocaine-prilocaine (EMLA) emulsion and effect of music distraction on the pain of intravenous cannulation. Pediatrics. 1994 May;93(5):797-801. PMID 8165081
- [Background] Bishai R, Taddio A, Bar-Oz B, Freedman MH, Koren G. Relative efficacy of amethocaine gel and lidocaine-prilocaine cream for Port-a-Cath puncture in children. Pediatrics. 1999 Sep;104(3):e31. doi: 10.1542/peds.104.3.e31. PMID 10469814
- [Background] Chen E, Zeltzer LK, Craske MG, Katz ER. Children's memories for painful cancer treatment procedures: implications for distress. Child Dev. 2000 Jul-Aug;71(4):933-47. doi: 10.1111/1467-8624.00200. PMID 11016557
- [Background] Cummings EA, Reid GJ, Finley AG, McGrath PJ, Ritchie JA. Prevalence and source of pain in pediatric inpatients. Pain. 1996 Nov;68(1):25-31. doi: 10.1016/S0304-3959(96)03163-6. PMID 9251995
- [Background] Eichenfield LF, Funk A, Fallon-Friedlander S, Cunningham BB. A clinical study to evaluate the efficacy of ELA-Max (4% liposomal lidocaine) as compared with eutectic mixture of local anesthetics cream for pain reduction of venipuncture in children. Pediatrics. 2002 Jun;109(6):1093-9. doi: 10.1542/peds.109.6.1093. PMID 12042548
- [Background] Fitzgerald M, Millard C, McIntosh N. Cutaneous hypersensitivity following peripheral tissue damage in newborn infants and its reversal with topical anaesthesia. Pain. 1989 Oct;39(1):31-36. doi: 10.1016/0304-3959(89)90172-3. PMID 2812853
- [Background] Halperin DL, Koren G, Attias D, Pellegrini E, Greenberg ML, Wyss M. Topical skin anesthesia for venous, subcutaneous drug reservoir and lumbar punctures in children. Pediatrics. 1989 Aug;84(2):281-4. PMID 2748256
- [Background] Humphrey GB, Boon CM, van Linden van den Heuvell GF, van de Wiel HB. The occurrence of high levels of acute behavioral distress in children and adolescents undergoing routine venipunctures. Pediatrics. 1992 Jul;90(1 Pt 1):87-91. PMID 1614786
- [Background] Kapelushnik J, Koren G, Solh H, Greenberg M, DeVeber L. Evaluating the efficacy of EMLA in alleviating pain associated with lumbar puncture; comparison of open and double-blinded protocols in children. Pain. 1990 Jul;42(1):31-34. doi: 10.1016/0304-3959(90)91088-Z. PMID 2234995
- [Background] Lawson RA, Smart NG, Gudgeon AC, Morton NS. Evaluation of an amethocaine gel preparation for percutaneous analgesia before venous cannulation in children. Br J Anaesth. 1995 Sep;75(3):282-5. doi: 10.1093/bja/75.3.282. PMID 7547043
- [Background] Ramsook C, Kozinetz CA, Moro-Sutherland D. Efficacy of ethyl chloride as a local anesthetic for venipuncture and intravenous cannula insertion in a pediatric emergency department. Pediatr Emerg Care. 2001 Oct;17(5):341-3. doi: 10.1097/00006565-200110000-00005. No abstract available. PMID 11673710
- [Background] Sethna NF, Verghese ST, Hannallah RS, Solodiuk JC, Zurakowski D, Berde CB. A randomized controlled trial to evaluate S-Caine patch for reducing pain associated with vascular access in children. Anesthesiology. 2005 Feb;102(2):403-8. doi: 10.1097/00000542-200502000-00025. PMID 15681958
- [Background] Wollin SR, Plummer JL, Owen H, Hawkins RM, Materazzo F, Morrison V. Anxiety in children having elective surgery. J Pediatr Nurs. 2004 Apr;19(2):128-32. doi: 10.1016/s0882-5963(03)00146-5. PMID 15077211
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children, ages 4 - 12 , who had outpatient clinic visits between June 2007 and August 2008 at an urban, tertiary care hospital and required venipunctures for medical care were recruited for this study.
Period: Overall Study
Arm/Group | EMLA Cream | Synera Patch
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EMLA Cream | Synera Patch | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.7 (2.5) | 8.9 (2.5) | 8.8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 21 | 19 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 7 | 4 | 11
  More than one race | 31 | 31 | 62
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100
Number of Participants with Prior Venipunctures [Number; unit: Participants] — Information about prior history of venipunctures was obtained from participants and participants' during initial interview.
  Participants
    Less than10 venipunctures | 29 | 27 | 56
    More than 10 venipunctures | 21 | 23 | 44
Number of participants with history of topical anesthetics use [Count of Participants; unit: Participants] — Information about prior use of topical anesthetics was obtained from participants and participants' during initial interview.
  Participants | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Participants Self-rating of Pain Using the Wong-Baker FACES Pain Rating Scale.
Description: Participants were asked to report their level of pain using a 6-point Wong-Baker FACES Pain Rating Scale ranging from 0, "no pain," to 5, "the most pain you can have." The Wong-Baker FACES Pain Rating Scale is a validated tool for measuring pain in patients as young as 3 years old. A FACES pain score less than or equal to 2 is considered no pain to mild pain, and is clinically acceptable. Studies have shown average FACES pain scores for children receiving vascular access with placebo to be 2.2 to 3.5.
Time Frame: immediately after completion of venipuncture
Measure: Count of Participants; unit: Participants
Arm/Group | EMLA Cream | Synera Patch
Number analyzed (Participants) | 50 | 50
Participants
  Participants with FACES Score = 0 (No pain) | 42 | 38
  Participants with FACES Score = 1 | 6 | 8
  Participants with FACES Score = 2 | 2 | 3
  Participants with FACES Score = 3 | 0 | 1
  Participants with FACES Score = 4 | 0 | 0
  Participants with FACES Score = 5 | 0 | 0

2. Secondary Outcome: Parent Rating of Child's Pain Using a 6-point NRS
Description: The Numerical Rating Scale (NRS) is a 6-point rating scale where 0= no pain and 5 = worst pain. Parents reported their own subjective evaluation of participants pain level. Each participant had only one parental assessment. Total number of parental assessment for each pain level on the 6-point NRS is reported as total number of participants experiencing that pain level.
Time Frame: immediately after venipuncture is completed
Population: Number of parent assessment for each pain level on the 6-point NRS. Each participant had only one parental assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | EMLA Cream | Synera Patch
Number analyzed (Participants) | 50 | 50
Participants
  number of participants with NRS=0 (no pain) | 42 | 41
  number of participants with NRS=1 | 6 | 5
  number of participants with NRS=2 | 1 | 1
  number of participants with NRS=3 | 1 | 2
  number of participants with NRS=4 | 0 | 0
  number of participants with NRS=5 | 0 | 1

3. Secondary Outcome: Blinded Observer's Subjective Ratings of Participants' Pain Level at Tourniquet Placement, Using a 6-point NRS
Description: The NRS (Numerical Rating Scale) is a 6-point rating scale where 0= no pain and 5 = worst pain. Blinded observers reported their own subjective evaluation of the level of pain experienced by the participants at tourniquet placement. Total number of participants subjectively evaluated as experiencing each pain level is reported.
Time Frame: before venipuncture
Measure: Count of Participants; unit: Participants
Arm/Group | EMLA Cream | Synera Patch
Number analyzed (Participants) | 50 | 50
Participants
  Participants evaluated at NRS = 0 (No pain) | 41 | 37
  Participants evaluated at NRS = 1 | 6 | 6
  Participants evaluated at NRS = 2 | 2 | 5
  Participants evaluated at NRS = 3 | 1 | 1
  Participants evaluated at NRS = 4 | 0 | 1
  Participants evaluated at NRS = 5 | 0 | 0

4. Secondary Outcome: Blinded Observer's Subjective Ratings of the Participant's Pain Level at Needle Insertion, Using a 6-point NRS
Description: The NRS (Numerical Rating Scale) is a 6-point rating scale where 0= no pain and 5 = worst pain. Blinded observers reported their own subjective evaluation of the level of pain experienced by the participants at needle insertion. Total number of participants subjectively evaluated as experiencing each pain level is reported.
Time Frame: during needle insertion
Measure: Count of Participants; unit: Participants
Arm/Group | EMLA Cream | Synera Patch
Number analyzed (Participants) | 50 | 50
Participants
  Participants evaluated at NRS = 0 (No pain) | 32 | 25
  Participants evaluated at NRS = 1 | 14 | 12
  Participants evaluated at NRS = 2 | 2 | 9
  Participants evaluated at NRS = 3 | 2 | 2
  Participants evaluated at NRS = 4 | 0 | 2
  Participants evaluated at NRS = 5 | 0 | 0

5. Secondary Outcome: Blinded Observer's Subjective Ratings of the Participant's Pain Level at 5 Minutes Post Venipuncture Procedure, Using a 6-point NRS
Description: The NRS (Numerical Rating Scale) is a 6-point rating scale where 0= no pain and 5 = worst pain. Blinded observers reported their own subjective evaluation of the level of pain participants were experiencing 5 minutes after the venipuncture was completed. Total number of participants subjectively evaluated as experiencing each pain level is reported.
Time Frame: 5 minutes post venipuncture
Measure: Count of Participants; unit: Participants
Arm/Group | EMLA Cream | Synera Patch
Number analyzed (Participants) | 50 | 50
Participants
  Participants evaluated at NRS = 0 (No pain) | 45 | 45
  Participants evaluated at NRS = 1 | 3 | 4
  Participants evaluated at NRS = 2 | 1 | 1
  Participants evaluated at NRS = 3 | 1 | 0
  Participants evaluated at NRS = 4 | 0 | 0
  Participants evaluated at NRS = 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Investigators monitored for adverse events during procedure and up to 20 minutes after removal of topical anesthetic.
Description: Skin reactions actively watched for during procedure. No major adverse outcomes, minor site reactions resolved shortly after removal of EMLA.
Arm/Group | EMLA Cream | Synera Patch
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 27/50 | 10/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMLA Cream (N=50) | Synera Patch (N=50)
Erythema (Skin and subcutaneous tissue disorders) | 6 | 7
Pruitis (Skin and subcutaneous tissue disorders) | 1 | 0
pallor (Skin and subcutaneous tissue disorders) | 20 | 3
Edema (Skin and subcutaneous tissue disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes